CLINICAL TRIAL: NCT04885478
Title: SARS-CoV-2 Infection Among Healthcare Professionals: Demographic Characteristics and Serological and Immune Responses Related to Progression's Phenotype (ProHEPiC-19)
Brief Title: Professional's Health in Epidemiological Crisis Covid-19
Acronym: ProHEpiC-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other); IrsiCaixa (Other); Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Pere Toran, MN, Family Physician, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: 4R20-105
Record Dates: First submitted 2021-05-12; First posted 2021-05-13 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; Serological test; Kinetics; T cell; Citokines
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Serum , plasma, nasopharyngeal swabs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy health care workers: ≥ 18 years of age
  Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki.
  To be a health care professional worker infected or exposed to SARS-CoV-2
  RT-PCR (SARS-CoV2), negative at baseline or follow up
  Anti-SARS-CoV-2 IgG and IgM antibodies (Nucleopcapside), negative positive at baseline or follow up
  Interventions: Other: Immune response monitoring , blood samples
- Infected health care workers: ≥ 18 years of age
  Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki.
  To be a health care professional worker infected or exposed to SARS-CoV-2
  RT-PCR (SARS-CoV2), positive at baseline or follow up
  Anti-SARS-CoV-2 IgG and IgM antibodies (Nucleopcapside), positive at baseline or follow up
  Interventions: Other: Immune response monitoring , blood samples

INTERVENTIONS:
Other: Immune response monitoring , blood samples — In both cohorts:
  -SARS-CoV-2 IgG and IgM antibodies, ( Nucleocapside, Spike) in 8 visits during a year.
  Infected HCW:
  * Cytokines and T-Cell determination at baseline, 30, 60,180 days, 365 after positive test ( RT-PCR or SARS-CoV-2 antibodies )
  * Covid-19 Symptoms, clinical monitoring

SUMMARY:
Introduction: Coronavirus Disease 2019 (COVID-19) has caused a global pandemic. Epidemiological and clinical inter-individual differences, symptomatology, recovery and humoral response against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) are key factors to better understand and predict the course of the pandemic. As Health Care Workers (HCWs) are caring for infected patients they are more susceptible to infection, which not only is critical for their own health but also because it results in a shortage of HCWs that seriously affects health services. Thus, maintaining the health and welfare of HCWs and enabling their rapid return to work is vital to overcome this crisis. The ProHEpiC-19 cohort presents data on the immune response of HCWs infected with SARS-CoV-2. This dynamic cohort was started in March 2020 and still continues including participants.

DETAILED DESCRIPTION:
Objectives:

Primary: To consolidate a prospective cohort of Health Care Workers (HCWs) to generate epidemiological and clinical high quality data. This information will be relevant to improve health policies and clinical COVID-19 protocols. This cohort will also be used as an ongoing platform to implement SARS-CoV-2 research projects with particular emphasis on incidence rate, reinfection, vaccines, and long term immune response.

Secondary:

1. To determine the kinetics of SARS-CoV-2 antibodies and cellular immune response in early, mid, and long periods of immunization.
2. To assess the relation between clinical variables and initial RT-PCR results with the interindividual differences in the immune response in early, mid, and long periods of immunization.
3. To analyze differentially expressed cytokines as biomarkers of disease progression in early, mid, and long periods of immunization.

Methods and analysis: Longitudinal, dynamic, prospective cohort study with a 12-month follow-up, which is being conducted in 4 primary-care centres and one hospital of Northern Metropolitana Nord of Barcelona (Spain). For now, the study consists of 1350 participants divided into 2 cohorts: 1) Healthy-Exposed HCWs: 675 not infected by SARS-CoV-2 (RT-PCR with a negative result and negative SARS-CoV-2 antibodies at baseline) and 2) Infected HCWs: 675 symptomatic participants (those with new persistent cough, temperature ≥37.5°C, anosmia, or ageusia or other compatible symptoms with COVID-19) or asymptomatic participants diagnosed by positive RT-PCR test and/or SARS-CoV-2 antibodies (IgM, IgG at baseline). Primary outcomes include: humoral and cellular immune response, quantitative antibodies to SARS-Cov-2, SARS-CoV-2 antibody levels related to progression phenotype, clinical spectrum of SARS-Cov-2, symptomatology, demographics and other variables that may be predictive of immune response.

Follow-up: baseline, 15 days, 1, 3, 6, 9 and 12 months. Findings to date: Current literature has shown that the immune response is maintained for a minimum of 2 months. Nevertheless little is known about the association between the immune response and the progression phenotype of COVID-19 .

Future plans: This prospective cohort offers the possibility to study associations between immune response and progression phenotype according to age and gender as well as long-term immune response. In turn, we will be able to examine possible cumulative effects, taking into account several clinical variables. The study is ongoing and we plan to extend it to increase the size of the cohort until 2024.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki.
* To be a health care professional worker infected or exposed to SARS-CoV-2.

Exclusion Criteria:

* < 18 years old
* Not to accept to take part in the study and/or not to sign the informed consent according to the Declaration of Helsinki.
* Not to be a health care professional worker exposed to SARS-CoV-2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter study (public primary care centers set in Mataró, Sabadell and Santa Perpètua and the public third level hospital Hospital Germans Tries i Pujol located in Badalona) with HCW cohorts recruited from Gerència Territorial Metropolitana Nord of the Catalan Institute of Health (ICS), which consists of 7,776 HCW, including physicians, nurses, COVID-19 researchers, medical residents and other essential workers in direct contact with patients during present and future pandemic waves.
Sampling Method: Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Creation prospective cohort of health care workers | Baseline, to 12 months after the beginning of the study
  Include 675 exposed HCW participants and 675 infected HCW participants againts SARS-CoV-2, cohorts will be compared at each time point in terms of sociodemographic, epidemiological, clinical, and immunological information available. an exploratory bivariate analysis will be performed using the tests of Chi Square, ANOVA, Kruskall-Walis, depending on the application conditions assumptions.
Cohort description demografics ( age, sex, academic level, housing characteristics, work variables ) | Baseline, to 12 months after the beginning of the study
  Descriptive analysis of the participants will be performed using the number and percentage for categorical variables, and mean and standard deviation or median and quartiles 1 and 3 for quantitative variables, an exploratory bivariate analysis will be performed using the tests of Chi Square, ANOVA, Kruskall-Walis, depending on the application conditions assumptions.
Cohort description clinical spectrum (asymptomatic, mild-moderate Illness, severe-critical) | Baseline, to 12 months after the beginning of the study
  Cohort comparison , an exploratory bivariate analysis will be performed using the tests of Chi Square, ANOVA, Kruskall-Walis, depending on the application conditions assumptions.

SECONDARY OUTCOMES:
Kinetics of SARS-CoV-2. IgM Nucleocapside | Baseline, 7 days, 15 days, 3, 6, 9 and 12 months after the beginning of the study
  IgM (nucleocapside) ELISA kits (Inmunodiagnostic Limited ©). Positivity thresholds were provided by the assay manufacturers and were considered positive with an index value greater than 1.1, indeterminate from 0.9 to 1.1 and negative if <0.9 index units
Kinetics of SARS-CoV-2. IgG Nucleocapside | Baseline, 7 days, 15 days, 3, 6, 9 and 12 months after the beginning of the study
  IgG (nucleocapside) ELISA kits (Inmunodiagnostic Limited ©). Positivity thresholds were provided by the assay manufacturers and were considered positive with an index value greater than 1.1, indeterminate from 0.9 to 1.1 and negative if <0.9 index units
Kinetics of SARS-CoV-2. IgG Spike | Baseline, 7 days, 15 days, 3, 6, 9 and 12 months after the beginning of the study
  IgG (spike). ELISA kits DECOV1901 (Demeditec Diagnostics GmbH©). Positivity thresholds were provided by the assay manufacturers and were considered positive with an index value greater than 40, indeterminate from 32 to 40 and negative if <32 Ul/ml
Kinetics of SARS-CoV-2. T-Cell | Baseline, 7 days, 15 days, 3, 6, 9 and 12 months after the beginning of the study
  SARS-CoV-2 specific CD4+ and CD8+ T-cell responses we performed an IFNγ ELISPOT assay. Wells will be considered positive if they contained at least 50 spot-forming cells per 106 PBMCs above the background level (2X mean + 3Xstandard deviation).
To assess the relation between clinical variables and initial RT-PCR results in the whole sample and by sex. | Baseline, to 12 months after the beginning of the study
  To study the differences between clinical spectrums and initial RT-PCR we will use ANOVAs or Kruskal-Wallis tests, after checking normality assumption using a Shapiro-test
To analyse the relation between clinical variables and the interindividual differences in the immune response in early, mid, and long periods of immunization in the whole sample and by sex | Baseline, 7 days, 15 days, 3, 6, 9 and 12 months after the beginning of the study
  To study the differences between clinical spectrums and immune response in early period we will use ANOVAs or Kruskal-Wallis tests, after checking normality assumption using a Shapiro-test . Similarly, to look for differences in antibody levels between sex, either a t-test or a Mann-Whitney test will be performed.
Cytokines as biomarkers of disease progression in early, mid, and long periods of immunization. | Baseline, 7 days, 15 days, 3, 6, 9 and 12 months after the beginning of the study
  Cryopreserved plasma samples will be used in a 45-plex assay of soluble mediators. The plates will be read with a Luminex instrument (Luminex 200, Austin Luminex, USA).Appropriate statistical tests (i.e. t-test or Mann-Whitney to compare between sexes and ANOVA or Kruskal-Wallis to compare between clinical spectrums) will be used after checking for normality (Shapiro-test)

CONTACTS AND LOCATIONS:
Overall Officials: Concepción Violán Fors, MD, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Jordi Gol i Gurina Foundation, Mataró, Barcelona, Spain

REFERENCES:
- [Background] Chen ZM, Fu JF, Shu Q, Chen YH, Hua CZ, Li FB, Lin R, Tang LF, Wang TL, Wang W, Wang YS, Xu WZ, Yang ZH, Ye S, Yuan TM, Zhang CM, Zhang YY. Diagnosis and treatment recommendations for pediatric respiratory infection caused by the 2019 novel coronavirus. World J Pediatr. 2020 Jun;16(3):240-246. doi: 10.1007/s12519-020-00345-5. Epub 2020 Feb 5. PMID 32026148
- [Background] Liu W, Fontanet A, Zhang PH, Zhan L, Xin ZT, Baril L, Tang F, Lv H, Cao WC. Two-year prospective study of the humoral immune response of patients with severe acute respiratory syndrome. J Infect Dis. 2006 Mar 15;193(6):792-5. doi: 10.1086/500469. Epub 2006 Feb 9. PMID 16479513
- [Background] Callow KA, Parry HF, Sergeant M, Tyrrell DA. The time course of the immune response to experimental coronavirus infection of man. Epidemiol Infect. 1990 Oct;105(2):435-46. doi: 10.1017/s0950268800048019. PMID 2170159
- [Result] Garcia-Sierra RM, Badia Perich E, Manresa Dominguez JM, Moreno Millan N, Sabate Cintas V, Romero Martinez M, Moreno Gabriel E, Pera G, Seda Gombau G, Montella Jordana N, Violan Fors C, Argerich Gonzalez MJ, Bonet Simo JM, Prat Gil N, Toran Monserrat P. [Descriptive study of the health service workers of a Primary Care Department confined by Covid-19.]. Rev Esp Salud Publica. 2020 Sep 3;94:e202009106. Spanish. PMID 32880381
- [Result] Huang AT, Garcia-Carreras B, Hitchings MDT, Yang B, Katzelnick LC, Rattigan SM, Borgert BA, Moreno CA, Solomon BD, Trimmer-Smith L, Etienne V, Rodriguez-Barraquer I, Lessler J, Salje H, Burke DS, Wesolowski A, Cummings DAT. A systematic review of antibody mediated immunity to coronaviruses: kinetics, correlates of protection, and association with severity. Nat Commun. 2020 Sep 17;11(1):4704. doi: 10.1038/s41467-020-18450-4. PMID 32943637
- [Derived] Violan C, Toran-Monserrat P, Quirant B, Lamonja-Vicente N, Carrasco-Ribelles LA, Chacon C, Manresa-Dominguez JM, Ramos-Roure F, Dacosta-Aguayo R, Palacios-Fernandez C, Roso-Llorach A, Pujol A, Ouchi D, Monteagudo M, Montero-Alia P, Garcia-Sierra R, Armestar F, Dolade M, Prat N, Bonet JM, Clotet B, Blanco I, Boigues-Pons M, Moreno-Millan N, Prado JG, Caceres EMM; ProHEpiC-19 study. Kinetics of humoral immune response over 17 months of COVID-19 pandemic in a large cohort of healthcare workers in Spain: the ProHEpiC-19 study. BMC Infect Dis. 2022 Sep 3;22(1):721. doi: 10.1186/s12879-022-07696-6. PMID 36057544

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT04885478/Prot_SAP_ICF_001.pdf